CLINICAL TRIAL: NCT06465927
Title: Clinical Significance of Appendicoliths in Elderly Patients Over 80 Years Old Undergoing Emergency Appendectomy: A Single-center Retrospective Study
Brief Title: Clinical Significance of Appendicoliths in Elderly Patients Over 80 Years Old Undergoing Emergency Appendectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhongshan-HHY-04
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Appendicoliths in Elderly Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical data collection — Clinical data of elderly acute appendicitis patients with an appendicolith who underwent emergency appendectomy were collected and analyzed.

SUMMARY:
Acute appendicitis with an appendicolith is one of the most common abdominal emergencies in elderly patients and is more likely to progress to gangrene and perforation. This study aimed to analyze the clinical data of patients over 80 years old who underwent emergency appendectomy for acute appendicitis, to explore the clinical significance of appendicoliths, and to improve treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who aged 80 years or older, who received conservative treatment for less than 24 hours before surgery, who had no peri-appendiceal abscess larger than 2 cm in diameter on CT scan, who underwent emergency appendectomy, and who had postoperative pathological confirmation of acute appendicitis.

Exclusion Criteria:

* Patients younger than 80 years, those with malignancies, and those with incomplete clinical or pathological records were excluded from the study.

Ages: 80 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The patients over 80 years old who underwent emergency appendectomy for acute appendicitis at the Department of Emergency Surgery of Zhongshan Hospital, Fudan University, from January 2016 to March 2023.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Morbidity of elderly patients undergoing emergency appendectomy | January 01, 2024 to December 31, 2024.
  Morbidity of elderly acute appendicitis patients with an appendicolith who underwent emergency appendectomy
Mortality of elderly patients undergoing emergency appendectomy | January 01, 2024 to December 31, 2024.
  Mortality of elderly acute appendicitis patients with an appendicolith who underwent emergency appendectomy